CLINICAL TRIAL: NCT00495235
Title: Case-Control Study of Insulin Resistance and Endometrial Cancer in Harris County, Texas
Brief Title: Study of Insulin Resistance and Endometrial Cancer in Harris County, Texas
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0164
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Polycystic Ovarian Syndrome; Insulin Resistance; Pre-diabetes; Harris County; PCOS; Uterus; Questionnaire; Body mass index; BMI
MeSH Terms: conditions — Endometrial Neoplasms; Polycystic Ovary Syndrome; Insulin Resistance; Glucose Intolerance | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample and, if diagnosed with endometrial cancer and had surgical removal of uterus, a piece of leftover tumor and surrounding normal tissue will be tested for markers of insulin resistance and PCOS.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Endometrial Cancer Group: Participants who have had endometrial cancer (cases).
  Interventions: Behavioral: Questionnaire
- Control Group: Participants who have not had endometrial cancer (controls).
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire taking about 20 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to find out if there is a link between insulin resistance (or pre-diabetes) and endometrial cancer.

Primary Objective:

1. To determine the association between insulin resistance and endometrial cancer in women in Harris County, Texas. 2. To assess the effect of body mass index (BMI) on the association between insulin resistance and endometrial cancer.

Secondary Objectives:

1. To explore the association between polycystic ovarian syndrome (PCOS) and endometrial cancer.
2. To assess the relationship between known reproductive risk factors, menstrual risk factors, family history and endometrial cancer.
3. To explore the molecular changes associated with insulin resistance and PCOS on normal endometrium and tumor tissue.

DETAILED DESCRIPTION:
This study will be comparing women who have had endometrial cancer (cases) to women who have not had endometrial cancer (controls) in Harris County, Texas to better understand the risk factors for getting endometrial cancer. Insulin resistance is a condition of pre-diabetes. Polycystic ovarian syndrome (PCOS) is a condition associated with irregular periods, obesity, infertility, and/or difficulty in getting pregnant. Both insulin resistance and PCOS are believed to increase a woman's risk of getting endometrial cancer.

As part of this study, you will be asked to fill out a questionnaire that asks about your medical history, weight history, family history, reproductive history, and birth control/hormone use. The questionnaire should take about 20 minutes to complete, and you will need to complete it only once. You will have your height and weight measured, and about 4 teaspoons of blood will be drawn to test for insulin resistance (or pre-diabetes). You will be required to fast, not eat or drink anything except water, for 8 hours before having this blood sample drawn. If you are premenopausal and still have both your ovaries, you will have an additional 4 teaspoons of blood drawn to test for PCOS. You will complete the questionnaire during your first visit or at home and will bring it back with you when you come back for your fasting blood test appointment.

If you have been diagnosed with endometrial cancer and have had surgery to remove your uterus, you will also be asked to give permission to use a piece of your leftover tumor and surrounding normal tissue to test for markers of insulin resistance and PCOS. This will be from tissue that was removed during your surgery and will not require another biopsy or surgery.

You will not be required to come back for any follow-up as part of this study. However, you will be asked to fill out a form that asks if you would be willing to be called in the future to participate in other studies.

This is an investigational study. A total of 700 women will take part in this multicenter study, 350 women with endometrial cancer and 350 women without endometrial cancer. A total of up to 350 women will be enrolled at M.D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histologically confirmed primary endometrial cancer, who will consent to be enrolled in the study no later than 12 weeks after their primary treatment. All stages, grades and histologic subtypes will be eligible.
2. Women who reside in Harris County, Texas. (Cases)
3. Patients must sign an informed consent for the study. (Cases)
4. Women must speak and understand English or Spanish. (Cases)
5. Women who reside in Harris County, Texas. (Controls)
6. No history of prior malignancy with the exception of non-melanoma skin cancer. (Controls)
7. Intact uterus. (Controls)
8. Patients must sign an informed consent for the study. (Controls)
9. Women must speak and understand English or Spanish. (Controls)

Exclusion Criteria:

1. Women who reside outside of Harris County, Texas. (Cases)
2. Patients unwilling or unable to provide informed consent. (Cases)
3. Metastatic cancer to the endometrium from a different primary. (Cases)
4. Women who do not speak and understand English or Spanish. (Cases)
5. Women who reside outside of Harris County, Texas. (Controls)
6. Previous hysterectomy. (Controls)
7. History of prior malignancy with the exception of non-melanoma skin cancer. (Controls)
8. Patients unwilling or unable to provide informed consent. (Controls)
9. Women who do not speak and understand English or Spanish. (Controls)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants from Harris County who have had endometrial cancer (cases) and those who have not (controls).
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2005-10; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Prevalence Rate of Insulin Resistance | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Karen H. Lu, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (8):
- United States (8):
  - Baylor College of Medicine/Clinics, Houston, Texas
  - Ben Taub Hospital, Houston, Texas
  - Gynecologic Oncology of Houston, Houston, Texas
  - Lyndon B. Johnson General Hospital, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org